CLINICAL TRIAL: NCT02955121
Title: IU Health Krannert Personalized Medicine Study - Influencing Prescriber Behavior for the Use of Clopidogrel
Brief Title: IU Health Krannert Personalized Medicine Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slower than anticipated recruitment
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Rolf Kreutz, MD. Associate Professor of Clinical Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1408765880
Record Dates: First submitted 2016-10-07; First posted 2016-11-04 (Estimated); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Coronary Artery Disease
Keywords: Cytochrome P-450 CYP2C19; Pharmacogenetics; Platelet Aggregation Inhibitors; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pharmacogenetic Results Available to Provider (Active Comparator): Genotyping for CYP2C19 variants is performed. The test results are integrated into the electronic health record and alerts are displayed to the prescriber. The ultimate decision regarding antiplatelet therapy is left to the prescriber
  Interventions: Other: Prescriber Access to Genetic Information
- Control Arm (No Intervention): No genotyping information is performed as part of clinical care. Standard therapy is followed. Genotyping will be performed at conclusion of study in control arm, and genotyping results will not be incorporated into electronic health record.

INTERVENTIONS:
Other: Prescriber Access to Genetic Information
  Arms: Pharmacogenetic Results Available to Provider

SUMMARY:
Randomized controlled study to examine physician use of pharmacogenetic information in patients receiving antiplatelet medication after percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
The study will randomize patients who have completed PCI and who are prescribed dual antiplatelet therapy to a genotype guided arm, in which CYP2C19 pharmacogenetic testing will be performed and a standard therapy arm without genetic testing. The study will examine the impact of pharmacogenetic testing on physician medication choice and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ischemic heart disease, who are prescribed dual antiplatelet therapy after percutaneous coronary intervention (PCI). Enrollment has to occur during index hospitalization or during outpatient visit for cath lab procedure.

Exclusion Criteria:

* Pregnant or breastfeeding.
* Unwilling or unable, in the opinion of the investigator, to comply with instructions on prescribed medicines.
* Prior known allergy or intolerance to clopidogrel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2016-11; Primary Completion 2019-08-09 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Change in prescription of antiplatelet therapy | one year
  Number of individuals whose initial P2Y12 inhibitor therapy was changed to another P2Y12 inhibitor during time of follow up

SECONDARY OUTCOMES:
Death, Myocardial Infarction, Stroke | one year
  Combined incidence of either death, myocardial infarction or stroke during follow up
Stent Thrombosis | one year
  Combined incidence of stent thrombosis according to Academic Research Consortium definitions during follow up
Urgent target vessel revascularization | one year
  Incidence of urgent target revascularization
Major and Minor Bleeding | one year
  Incidence of Major or Minor Bleeding according to GUSTO criteria during follow up

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Kreutz, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Health Methodist Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified Data Sharing only